CLINICAL TRIAL: NCT07076485
Title: Shortening Adjuvant Photon and Proton Irradiation (SAPPHIRe-II): A 4 Cohort, Randomized, Phase II Multi-center Trial Evaluating Shorter Schedules of Adjuvant Regional Nodal Irradiation Among Women and Men With Node-positive and High-risk Node-negative Invasive Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0779; NCI-2025-05190 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-07-15; First posted 2025-07-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- High-Risk Lumpectomy Cohort Arm 1: Moderately Hypofractionated Breast+RNI with SIB (Experimental)
  Interventions: Radiation: Moderately Hypofractionated Radiation
- High-Risk Lumpectomy Cohort Arm 2: Moderately Hypofractionated Breast+RNI with Sequential Boost (Other)
  Interventions: Radiation: Moderately Hypofractionated Radiation
- High-Risk Mastectomy Cohort Arm 1: Moderately Hypofractionated Chest Wall+RNI with SIB (Experimental)
  Interventions: Radiation: Moderately Hypofractionated Radiation
- High-Risk Mastectomy Cohort Arm 2: Moderately Hypofractionated Chest Wall+RNI with Sequential Boost (Other)
  Interventions: Radiation: Moderately Hypofractionated Radiation
- Low-Risk Lumpectomy Cohort Arm 1: Ultrahypofractionated Breast+RNI with SIB (Experimental)
  Interventions: Radiation: Ultrahypofractionated Radiation
- Low-Risk Lumpectomy Cohort Arm 2: Moderately Hypofractionated Breast+RNI with SIB (Other)
  Interventions: Radiation: Moderately Hypofractionated Radiation
- Low-Risk Mastectomy Cohort Arm 1: Ultrahypofractionated Chest Wall+RNI (Experimental)
  Interventions: Radiation: Ultrahypofractionated Radiation
- Low-Risk Mastectomy Cohort Arm 2: Moderately Hypofractionated Breast+RNI (Other)
  Interventions: Radiation: Moderately Hypofractionated Radiation

INTERVENTIONS:
Radiation: Ultrahypofractionated Radiation — Given by infusion
  Arms: Low-Risk Lumpectomy Cohort Arm 1: Ultrahypofractionated Breast+RNI with SIB; Low-Risk Mastectomy Cohort Arm 1: Ultrahypofractionated Chest Wall+RNI
Radiation: Moderately Hypofractionated Radiation — Given by infusion
  Arms: High-Risk Lumpectomy Cohort Arm 1: Moderately Hypofractionated Breast+RNI with SIB; High-Risk Lumpectomy Cohort Arm 2: Moderately Hypofractionated Breast+RNI with Sequential Boost; High-Risk Mastectomy Cohort Arm 1: Moderately Hypofractionated Chest Wall+RNI with SIB; High-Risk Mastectomy Cohort Arm 2: Moderately Hypofractionated Chest Wall+RNI with Sequential Boost; Low-Risk Lumpectomy Cohort Arm 2: Moderately Hypofractionated Breast+RNI with SIB; Low-Risk Mastectomy Cohort Arm 2: Moderately Hypofractionated Breast+RNI

SUMMARY:
To learn about the effects of shorter RNI regimens in patients with breast cance who have had a lumpectomy or mastectomy and who are at higher risk for lower risk for the disease returning.

DETAILED DESCRIPTION:
Primary Objective:

To compare the occurrence of any grade 2 or higher NCI CTCAE toxicity from start of RNI through 18 months follow up by treatment arm for each of the four randomized cohorts (low-risk lumpectomy, low-risk mastectomy, high-risk lumpectomy, high-risk mastectomy).

Secondary Objectives:

To compare treatment toxicity, local-regional control, disease-free survival, and overall survival by treatment arm for each of the four randomized cohorts.

To compare patient-reported outcomes including cosmetic satisfaction, physical wellbeing, lymphatic function, and financial toxicity by treatment arm for each of the four randomized cohorts.

To compare photographic outcome of the treated breast or reconstructed breast by treatment arm for each of the four randomized cohorts.

To evaluate and compare radiation treatment plans by treatment arm for each of the four randomized cohorts, including target coverage, dose to organs at risk, dose homogeneity, and low-dose scatter.

To compare biometric data before, during, and after radiation collected by patients' personal Apple Watches.

ELIGIBILITY:
Inclusion Criteria:

Eligibility Criteria Applicable to All Cohorts

Histologically confirmed invasive breast cancer (nodal involvement from presumed invasive breast cancer in the setting of occult breast cancer is sufficient to meet this criteria)

1. Regional nodal irradiation recommended by treating radiation oncologist. 2 Negative final surgical margins. 3 No more than 12 weeks have elapsed since final breast/lymph node surgery for patients treated with surgery alone or neoadjuvant chemotherapy. No more than 12 weeks have elapsed since final cytotoxic chemotherapy for patients who received adjuvant chemotherapy. 5. Age ≥18 years. Because breast cancer is exceedingly rare in patients < 18 years of age, children are excluded from this study. 6. Patients with a prior or concurrent malignancy are eligible provided that the natural history and treatment of the prior or concurrent malignancy does not interfere with the safety or efficacy assessment of the investigational radiation regimen used in this trial. 7. Ability to understand and the willingness to sign a written informed consent document. 8. Concurrent enrollment on other observational, translational, or therapeutic studies is allowed provided there is no direct conflict between the other protocol and the radiation regimen proscribed in this trial.

Eligibility Criteria for the Low-Risk Lumpectomy Cohort

1. For patients treated with upfront surgery, pathologic stage pT0-T4b N0-N3a breast cancer without infraclavicular or internal mammary nodal involvement.
2. For patients treated with neoadjuvant chemotherapy, clinical stage cT0-T4b N0-N2a breast cancer.
3. Treated with lumpectomy (or axillary surgery only in the case of occult primary breast cancer)
4. No nodal boost recommended by the treating radiation oncologist.

Eligibility Criteria for the High-Risk Lumpectomy Cohort

1. Treated with neoadjuvant chemotherapy
2. Clinical stage cT0-T4b N1-N3a/b/c
3. Treated with lumpectomy (or axillary surgery only in the case of occult primary breast cancer)
4. Nodal boost recommended by the treating radiation oncologist.

Eligibility Criteria for the Low-Risk Mastectomy Cohort

1. For patients treated with upfront surgery, pathologic stage T0-T2 N0-N2a
2. For patients treated with neoadjuvant chemotherapy, clinical stage T0-T3 N0- N2a
3. For patients treated with neoadjuvant chemotherapy, residual cellularity of primary tumor ≤ 20%.
4. Treated with mastectomy
5. Negative surgical margins ≥ 2 mm.
6. No or only focal lymphovascular space invasion.
7. Age ≥ 40 years
8. Chest wall boost NOT recommended by treating radiation oncologist.

Eligibility Criteria for High-Risk Mastectomy Cohort

1. For patients treated with upfront surgery, pathologic stage T0-T4d N0-N3c
2. For patients treated with neoadjuvant chemotherapy, clinical stage T0-T4d N0- N3c
3. Treated with mastectomy
4. Chest wall boost and/or nodal boost recommended by treating radiation oncologist

Pregnancy Status (applicable to all cohorts)

Therapeutic radiation is known to be teratogenic. As a result, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of radiation treatment. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

* Postmenopausal (no menses in greater than or equal to 12 consecutive months).
* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure.

Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the radiation therapy course is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Men treated or enrolled on this protocol must also agree to use adequate contraception during the radiation treatment course.

Pregnancy testing at the time of study enrollment is not required of women who enroll. However, all patients must comply with the Institutional Pregnancy Assessment Policy (# CLN1114) which requires pregnancy testing within 7 days prior to simulation.

Exclusion Criteria:

History of therapeutic radiation overlapping with the index breast or nodal basins that require radiation therapy.

History of scleroderma

Pregnant women are excluded from this study because ionizing radiation has the potential for teratogenic or abortifacient effects.

Patients with psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Smith, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org